CLINICAL TRIAL: NCT03028103
Title: An Open-Label, Multicenter, Two-Part, Phase 1 Study to Characterize the Effects of a Moderate CYP3A Inhibitor on the Pharmacokinetics of Tazemetostat (EPZ-6438) (Part A), the Effects of Tazemetostat on the Pharmacokinetics of CYP2C8 and CYP2C19 Substrates, and the Effect of Increased Gastric pH on the Pharmacokinetics of Tazemetostat (Part B) in Subjects With B-cell Lymphoma or Advanced Solid Tumors
Brief Title: Open-Label, Multicenter, Two-Part, Phase 1 Study to Characterize Effects of a Moderate CYP3A Inhibitor on PK of Tazemetostat, Effects of Tazemetostat on PK of CYP2C8 and CYP2C19 Substrates, and Effect of Increased Gastric pH on PK of Tazemetostat in B-cell Lymphoma or Advanced Solid Tumor Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Epizyme, Inc. (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EZH-105
Record Dates: First submitted 2016-12-19; First posted 2017-01-23 (Estimated); Results first posted 2021-04-19 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Diffuse Large B Cell Lymphoma; Primary Mediastinal Lymphoma; Mantle Cell Lymphoma; Advanced Solid Tumor; Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — tazemetostat; Fluconazole; Omeprazole; repaglinide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Part A and B (Experimental): Part A: Subjects enrolled in Part A will receive treatment with oral tazemetostat tablets 400 mg BID for 24 days beginning on Day 1. Subjects will receive fluconazole 400 mg once daily for 4 days starting on Day 16. Tazemetostat 400 mg BID will continue through Day 24. Subjects will then receive tazemetostat 800 mg BID starting on Day 25.
  Part B: Subjects enrolled in Part B will receive single oral doses of repaglinide 0.25 mg and omeprazole 20 mg on Day 1. Administration of tazemetostat 800 mg BID will begin on Day 2. On Day 16, subjects again will receive single oral doses of repaglinide 0.25 mg and omeprazole 20 mg approximately 1 hour after the morning dose of tazemetostat. Subjects also will receive omeprazole 20 mg once daily in the morning on Days 16 through 19.
  Interventions: Drug: Tazemetostat; Drug: Fluconazole; Drug: Omeprazole; Drug: Repaglinide

INTERVENTIONS:
Drug: Tazemetostat — Tazemetostat is a selective oral small molecule inhibitor of EZH2
  Other Names: EPZ-6438, E7438
Drug: Fluconazole — 200mg will be orally administered QD for 4 days in order to determine CYP3A4 inhibition when administered concomitantly with tazemetostat
Drug: Omeprazole — Using omeprazole as a probe substrate, 20mg will be orally administered for a total of 5 days in order to determine the potential of tazemetostat to inhibit or induce CYP2C19. Omeprazole is also being used to determine the effect of increased gastric pH on metabolism of tazemetostat.
Drug: Repaglinide — Using repaglinide as a probe substrate, 25mg will be orally administered for a total of 2 days in order to determine the potential of tazemetostat to inhibit or induce CYP2C8.

SUMMARY:
This is a Phase 1, open-label, two-part, safety, PK, and activity study designed to characterize the DDI potential of tazemetostat. Tazemetostat will be taken orally BID continuously in 28-day cycles in both study parts.

ELIGIBILITY:
Inclusion criteria

1. Male or female ≥ 18 years of age at time of consent
2. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
3. Has the ability to understand informed consent and provided signed written informed consent

   Must meet one of the following criteria:
4. Has histologically confirmed diffuse large B-cell lymphoma (DLBCL), primary mediastinal B-cell lymphoma (PMBCL), marginal zone lymphoma (MZL), mantle cell lymphoma (MCL) and have relapsed or refractory disease following at least two lines of prior standard therapy, including alkylator/anthracycline (unless anthracycline-based chemotherapy is contraindicated)/anti-CD20-based therapy (R-CHOP; rituximab, doxorubicin, cyclophosphamide, vincristine, and prednisolone or prednisone, or equivalent) AND must be considered unable to benefit from intensification treatment with autologous hematopoietic stem cell transplantation (ASCT), as defined by meeting at least one of the following criteria:

   1. Relapsed following, or refractory to, previous ASCT
   2. Did not achieve at least a partial response (PR) to a standard salvage regimen (e.g., R-ICE; rituximab, ifosfamide, carboplatin, etoposide, or R-DHAP; rituximab, dexamethasone, cytarabine, cisplatin)
   3. Ineligible for intensification treatment due to age or significant comorbidity
   4. Ineligible for intensification treatment due to failure to mobilize an acceptable number of hematopoietic stem cells
   5. Refused intensification treatment and/or ASCT Note: Subjects with prior radiotherapy will be included; however, radiotherapy alone will not be considered a separate systemic treatment regimen.

   Note: Subjects with prior radiotherapy will be included; however, radiotherapy alone will not be considered a separate systemic treatment regimen.

   OR
5. Has histologically confirmed FL, all grades. Subjects must have relapsed/refractory disease following at least 2 standard lines of systemic therapy, including at least 1 anti-CD20-based regimen (eg, rituximab), as well as alkalating agents (eg, cyclophosphamide or bendamustine), and have no curative option with other available therapies OR have a contra-indication to their use. Subjects with prior ASCT may be included. Transformed disease is permitted.

   Note: Subjects with prior radiotherapy will be included; however, radiotherapy alone will not be considered a separate systemic treatment regimen.

   OR
6. Histologically and/or cytologically confirmed advanced or metastatic solid tumor that has progressed after treatment with approved therapies or for which there are no standard therapies available
7. Must have evaluable or measurable disease
8. Has all prior treatment (i.e., chemotherapy, immunotherapy, radiotherapy) related clinically significant toxicities resolve to ≤ Grade 1 per NCI CTCAE, Version 4.03 or are clinically stable and not clinically significant, at time of consent
9. Time required between the last dose of the latest therapy and the first dose of study drug:

   1. Chemotherapy: cytotoxic At least 21 days
   2. Chemotherapy: nitrosoureas At least 6 weeks
   3. Chemotherapy: non-cytotoxic (e.g., small molecule inhibitor) At least 14 days
   4. Monoclonal antibody (ies) At least 28 days
   5. Non-antibody immunotherapy (e.g., tumor vaccine) At least 42 days
   6. At least 14 days for stereotactic radiosurgery
   7. At least 12 weeks for craniospinal, ≥50% radiation of pelvis, or total body irradiation prior to first dose of study drug
   8. Autologous hematopoietic cell infusion after high dose therapy At least 60 days
   9. Hematopoietic growth factor At least 14 days
10. Has adequate hematologic (bone marrow [BM] and coagulation factors), renal and hepatic function

    1. Hemoglobin ≥9 g/dL
    2. Platelets ≥75,000/mm3 (≥75 × 10^9/L)
    3. ANC: for patients with lymphoma ≥750/mm3 (≥0.75 × 10^9/L), for patients with advanced solid tumors ≥1,000/mm3 (≥1.0 × 10^9/L),
    4. PT <1.5 ULN
    5. PTT <1.5 ULN
    6. eGFR ≥ 50 mL/min/1.73 m2
    7. Conjugated bilirubin <1.5 × ULN
    8. AST <3 × ULN
    9. ALT <3 × ULN

    NOTE: Laboratory results obtained during screening should be used to determine eligibility criteria. In situations where laboratory results are outside the permitted range, the investigator may retest the subject and the subsequent within range screening result may be used to determine the subject's eligibility.
11. Has a QT interval corrected by Fridericia's formula (QTcF) ≤480 msec
12. Subjects with a history of Hepatitis B or C are eligible on the condition that subjects have adequate liver function as defined by the protocol and are hepatitis B surface antigen negative and/or have undetectable HCV RNA.
13. Male subjects must refrain from donating sperm starting at the planned first dose of investigational product (IP) until 30 days following the last dose of IP
14. Male subjects with a female partner of childbearing potential must:

    1. Be vasectomized, or
    2. Remain abstinent or use a condom as defined in Section 8.3.8.4.2, starting at the planned first dose of IP until 30 days following the last dose of IP. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, sympto-thermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception.
15. Female partners of male subjects who are of childbearing potential must also adhere to one of the following:

    1. Placement of an intrauterine device or intrauterine system.
    2. Established use of oral, injected, or implanted hormonal methods of contraception or use of a barrier method of contraception.
    3. Progesterone only oral contraception, where inhibition of ovulation is not the primary mode of action.
16. Women of childbearing potential or female partners of male subjects must abide by the contraception measures defined by the protocol

Exclusion criteria:

1. Is pregnant or nursing
2. Has active central nervous system (CNS) or leptomeningeal metastasis
3. Has had a prior malignancy other than the malignancies under study Exception: Subject who has been disease-free for 3 years, or a subject with a history of a completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
4. Has thrombocytopenia, neutropenia, or anemia of Grade ≥3 (per CTCAE 4.03 criteria) and any prior history of myeloid malignancies, including myelodysplastic syndrome (MDS).

   NOTE: Bone marrow aspirate/biopsy will be conducted following abnormal peripheral blood smear morphology assessment conducted by the local laboratory. Cytogenetic testing and DNA sequencing will be conducted following an abnormal result of bone marrow aspirate/biopsy.
5. Has a prior history of T-LBL/T-ALL.
6. Has had major surgery within 3 weeks prior to enrollment NOTE: Minor surgery (e.g., minor biopsy, central venous catheter placement) is permitted within 3 weeks prior to enrollment.
7. Is unwilling to exclude grapefruit juice, Seville oranges, and grapefruit from the diet and all foods that contain those fruits from time of enrollment to while on study
8. Has cardiovascular impairment, history of congestive heart failure greater than NYHA Class II uncontrolled arterial hypertension, unstable angina, myocardial infarction, or stroke within 6 months prior to the planned first dose of tazemetostat; or ventricular cardiac arrhythmia requiring medical treatment
9. Subjects taking medications that are known potent or moderate inducers/ inhibitors of CYP3A4 (including St. John's Wort)
10. Has an active infection or recent history (<30 days before study drug administration) requiring systemic treatment
11. Is immunocompromised, including subjects with known human immunodeficiency virus (HIV) infection
12. Has known hypersensitivity to any of the components of IP.
13. Is unable to take oral medications, has a history of surgery that would interfere with the administration or absorption of oral medication, has malabsorption syndrome or any other uncontrolled gastrointestinal condition (e.g., nausea, diarrhea or vomiting) that might impair the bioavailability of IP
14. Has an uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, or psychiatric illness/social situations that would limit compliance with study requirements.
15. Is unwilling to adhere to contraception criteria from time of enrollment in study to at least 30 days after last dose of IP.
16. A history of bleeding (i.e., hemoptysis, hematuria, gastrointestinal blood loss, epistaxis, or others with greater than Grade 1 according to NCI CTCAE Version 4.03) within 1 month prior to beginning therapy or any clinical indications of current active bleeding.
17. Clinical history, current alcohol (ethanol), or illicit drug use which, in the judgment of the investigator, will interfere with the subject's ability to comply with the dosing schedule and protocol-specified evaluations.
18. Regular alcohol consumption averaging more than seven drinks/week for women and 14 drinks/week for men within 6 months of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-11-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Arizona Cancer Center, Tucson, Arizona
  - Moffitt Cancer Center, Tampa, Florida
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Subjects enrolled in Part A received treatment with oral tazemetostat tablets 400 mg twice daily for 24 days beginning on Day 1. Blood samples for the analysis of plasma tazemetostat and its metabolites concentrations were collected predose and over 8 hours after the morning dose of tazemetostat on Day 15. Subjects received fluconazole 400 mg once daily for 4 days starting on Day 16. On Day 19, blood samples for the analysis of plasma tazemetostat, its metabolites, and fluconazole were collected predose and over 8 hours after the morning tazemetostat dose. Tazemetostat 400 mg twice daily continued through Day 24. Subjects then received tazemetostat 800 mg twice daily starting on Day 25.
- Part B: Subjects enrolled in Part B received single oral doses of repaglinide 0.25 mg and omeprazole 20 mg on Day 1. Administration of tazemetostat 800 mg twice daily began on Day 2. On Day 16, subjects again received single oral doses of repaglinide 0.25 mg and omeprazole 20 mg approximately 1 hour after the morning dose of tazemetostat. Subjects also received omeprazole 20 mg once daily in the morning on Days 16 through 19. Blood samples for analysis of plasma repaglinide, repaglinide metabolites, omeprazole, 5-OH-omeprazole, and omeprazole sulfone were collected predose and over 7 hours after administration on Day 1 and Day 16. Blood samples for analysis of plasma tazemetostat and metabolites were collected over 8 hours after administration of the morning dose on Day 16 and Day 19.
Period: Overall Study
Arm/Group | Part A | Part B
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A | Part B | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 11 | 20
  >=65 years | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.9 (15.10) | 48.8 (17.75) | 55.8 (17.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 6 | 9 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 15 | 13 | 28
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 14 | 12 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 16 | 32
Baseline Disease Characteristics and Prior Therapies [Count of Participants; unit: Participants]
  Lymphoma | 10 | 3 | 13
  Advanced Solid tumors | 6 | 13 | 19
  Stage at diagnosis: I | 0 | 0 | 0
  Stage at diagnosis: II | 1 | 1 | 2
  Stage at diagnosis: III | 5 | 3 | 8
  Stage at diagnosis: IV | 8 | 10 | 18
  Stage at diagnosis: Unknown | 2 | 2 | 4
  Progressive disease prior to study entry | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Part A: Effect of CYP3A Inhibition by Fluconazole on the PK of Tazemetostat (AUC0-t, AUC0-8)
Time Frame: Days 15 and 19, 0 to 8 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Part A: Part A: Subjects enrolled in Part A will receive treatment with oral tazemetostat tablets 400 mg BID for 24 days beginning on Day 1. Subjects will receive fluconazole 400 mg once daily for 4 days starting on Day 16. Tazemetostat 400 mg BID will continue through Day 24. Subjects will then receive tazemetostat 800 mg BID starting on Day 25.
Arm/Group | Part A
Number analyzed (Participants) | 14
h*ng/mL
  Part: A; Day 15; Treatment: Tazemetostat Alone; Analyte: EPZ-6438 | 1340 (1180)
  Part: A; Day 19; Treatment: Tazemetostat with Fluconazole; Analyte: EPZ-6438 | 4100 (2680)

2. Primary Outcome: Part A: Cmax of Tazemetostat During Co-administration With Fluconazole
Time Frame: Days 15 and 19, 0 to 8 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A
Number analyzed (Participants) | 14
ng/mL
  Part: A; Day 15; Treatment: Tazemetostat Alone; Analyte: EPZ-6438 | 426 (337)
  Part: A; Day 19; Treatment: Tazemetostat with Fluconazole; Analyte: EPZ-6438 | 968 (801)

3. Primary Outcome: Part B: The Potential of Tazemetostat to Inhibit or Induce CYP2C8 Using Repaglinide as a Probe Substrate (AUC0-t, AUC0-∞)
Time Frame: Days 1 and 16, 0 to 8 hours post-dose
Population: In Part B, 13 subjects completed taking omeprazole and repaglinide on Day 1, with tazemetostat on Day 16 and 11 subjects completed taking tazemetostat alone on Day 19.
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Part B: Part B: Subjects enrolled in Part B will receive single oral doses of repaglinide 0.25 mg and omeprazole 20 mg on Day 1. Administration of tazemetostat 800 mg BID will begin on Day 2. On Day 16, subjects again will receive single oral doses of repaglinide 0.25 mg and omeprazole 20 mg approximately 1 hour after the morning dose of tazemetostat. Subjects also will receive omeprazole 20 mg once daily in the morning on Days 16 through 19.
Arm/Group | Part B
Number analyzed (Participants) | 13
h*ng/mL
  Part: B; Day 1; Treatment: Repaglinide Alone; Analyte: Repaglinide - AUC(0-t) | 8.16 (13.7)
  Part: B; Day 16; Treatment: Repaglinide with Tazemetostat; Analyte: Repaglinide - AUC(0-t) | 14.7 (15.1)
  Part: B; Day 1; Treatment: Repaglinide Alone; Analyte: Repaglinide - AUC(0-∞) | 12.7 (19.4)
  Part: B; Day 16; Treatment: Repaglinide with Tazemetostat; Analyte: Repaglinide - AUC(0-∞) | 17 (15.7)

4. Primary Outcome: Part B: Cmax of Repaglinide During Co-administration With Tazemetostat
Time Frame: Days 1 and 16, 0 to 8 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B
Number analyzed (Participants) | 13
ng/mL
  Part: B; Day 1; Treatment: Repaglinide Alone; Analyte: Repaglinide | 5.14 (8.28)
  Part: B; Day 16; Treatment: Repaglinide with Tazemetostat; Analyte: Repaglinide | 7.75 (8.73)

5. Primary Outcome: Part B: The Potential of Tazemetostat to Inhibit or Induce CYP2C19 Using Omeprazole as Probe a Substrate (AUC0-t, AUC0-∞)
Time Frame: Days 1 and 16, 0 to 8 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part B
Number analyzed (Participants) | 13
h*ng/mL
  Part: B; Day 1; Treatment: Omeprazole Alone; Analyte: Omeprazole - AUC(0-t) | 600 (1600)
  Part: B; Day 16; Treatment: Omeprazole with Tazemetostat; Analyte: Omeprazole - AUC(0-t) | 480 (837)
  Part: B; Day 1; Treatment: Omeprazole Alone; Analyte: Omeprazole - AUC(0-∞) | 672 (463)
  Part: B; Day 16; Treatment: Omeprazole with Tazemetostat; Analyte: Omeprazole - AUC(0-∞) | 1120 (1530)

6. Primary Outcome: Part B: Cmax of Omeprazole During Co-administration With Tazemetostat
Time Frame: Days 1 and 16, 0 to 8 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B
Number analyzed (Participants) | 13
ng/mL
  Part: B; Day 1; Treatment: Omeprazole Alone; Analyte: Omeprazole | 253 (462)
  Part: B; Day 16; Treatment: Omeprazole with Tazemetostat; Analyte: Omeprazole | 207 (275)

7. Primary Outcome: Part B: Effect of Increased Gastric pH by Omeprazole on the PK of Tazemetostat (AUC0-t, AUC0-8)
Time Frame: Days 16 and 19, 0 to 8 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part B
Number analyzed (Participants) | 13
h*ng/mL
  Part: B; Day 16; Treatment: Omeprazole with Tazemetostat; Analyte: EPZ-6438 - AUC(0-t) | 1780 (2010)
  Part: B; Day 19; Treatment: Tazemetostat Alone; Analyte: EPZ-6438 - AUC(0-t): number analyzed (Participants) | 11
  Part: B; Day 19; Treatment: Tazemetostat Alone; Analyte: EPZ-6438 - AUC(0-t) | 2150 (1030)

8. Primary Outcome: Part B: Cmax of Tazemetostat During Co-administration With Omeprazole
Time Frame: Days 16 and 19, 0 to 8 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B
Number analyzed (Participants) | 13
ng/mL
  Part: B; Day 16; Treatment: Omeprazole with Tazemetostat; Analyte: EPZ-6438 | 521 (627)
  Part: B; Day 19; Treatment: Tazemetostat Alone; Analyte: EPZ-6438: number analyzed (Participants) | 11
  Part: B; Day 19; Treatment: Tazemetostat Alone; Analyte: EPZ-6438 | 641 (404)

9. Secondary Outcome: Incidence of Treatment-emergent Adverse Events as a Measure of Safety
Time Frame: From the first dose of study treatment until the earlier of either 30 days after the discontinuation of study treatment or until the initiation of subsequent anticancer therapy, up to 2 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A | Part B
Number analyzed (Participants) | 16 | 16
Participants
  Any TEAE | 12 | 14
  Any TEAE Grade 3 or 4 | 7 | 8
  Any Treatment-Related TEAE | 9 | 10
  Any Treatment-Related TEAE Grade 3 or 4 | 4 | 3
  Any TEAE Leading to Dose Reduction | 2 | 2
  Any TEAE Leading to Study Drug Interruption | 3 | 6
  Any TEAE Leading to Study Drug Discontinuation | 0 | 0
  Any TESAE | 4 | 6
  Any Treatment-Related TESAE | 1 | 0
  Any Protocol Defined AE of Special Interest | 0 | 0

10. Secondary Outcome: Part A: PK of Tazemetostat and Its Metabolites After Administration Alone and With Fluconazole (AUC0-t, AUC0-8)
Time Frame: Days 15 and 19, 0 to 8 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part A
Number analyzed (Participants) | 14
h*ng/mL
  Part: A; Day 15; Treatment: Tazemetostat Alone; Analyte: EPZ-6930 (ER-897387) | 2590 (1200)
  Part: A; Day 19; Treatment: Tazemetostat with Fluconazole; Analyte: EPZ-6930 (ER-897387) | 2860 (1600)
  Part: A; Day 15; Treatment: Tazemetostat Alone; Analyte: EPZ006931 | 770 (630)
  Part: A; Day 19; Treatment: Tazemetostat with Fluconazole; Analyte: EPZ006931 | 921 (780)
  Part: A; Day 15; Treatment: Tazemetostat Alone; Analyte: EPZ034163 | 276 (415)
  Part: A; Day 19; Treatment: Tazemetostat with Fluconazole; Analyte: EPZ034163 | 295 (430)

11. Secondary Outcome: Part A: Tmax of Tazemetostat After Administration Alone and With Fluconazole
Time Frame: Days 15 and 19, 0 to 8 hours post-dose
Measure: Median (Standard Deviation); unit: hours
Arm/Group | Part A
Number analyzed (Participants) | 14
hours
  Part: A; Day 15; Treatment: Tazemetostat Alone; Analyte: EPZ-6438 | 1.13 (0.87)
  Part: A; Day 19; Treatment: Tazemetostat with Fluconazole; Analyte: EPZ-6438 | 2 (0.84)

12. Secondary Outcome: Part A: t1/2 of Tazemetostat After Administration Alone and With Fluconazole
Time Frame: Days 15 and 19, 0 to 8 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: hours
Arm/Group | Part A
Number analyzed (Participants) | 14
hours
  Part: A; Day 15; Treatment: Tazemetostat Alone; Analyte: EPZ-6438 | 2.88 (0.491)
  Part: A; Day 19; Treatment: Tazemetostat with Fluconazole; Analyte: EPZ-6438 | 3.56 (0.453)

13. Secondary Outcome: Part A: Cmax of Tazemetostat Metabolites After Administration Alone and With Fluconazole
Time Frame: Days 15 and 19, 0 to 8 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A
Number analyzed (Participants) | 14
ng/mL
  Part: A; Day 15; Treatment: Tazemetostat Alone; Analyte: EPZ-6930 (ER-897387) | 629 (270)
  Part: A; Day 19; Treatment: Tazemetostat with Fluconazole; Analyte: EPZ-6930 (ER-897387) | 548 (288)
  Part: A; Day 15; Treatment: Tazemetostat Alone; Analyte: EPZ006931 | 166 (105)
  Part: A; Day 19; Treatment: Tazemetostat with Fluconazole; Analyte: EPZ006931 | 167 (153)
  Part: A; Day 15; Treatment: Tazemetostat Alone; Analyte: EPZ034163 | 46 (56.7)
  Part: A; Day 19; Treatment: Tazemetostat with Fluconazole; Analyte: EPZ034163 | 47.1 (61.4)

14. Secondary Outcome: Part A: Tmax of Tazemetostat Metabolites After Administration Alone and With Fluconazole
Time Frame: Days 15 and 19, 0 to 8 hours post-dose
Measure: Median (Standard Deviation); unit: hours
Arm/Group | Part A
Number analyzed (Participants) | 14
hours
  Part: A; Day 15; Treatment: Tazemetostat Alone; Analyte: EPZ-6930 (ER-897387) | 2.01 (0.65)
  Part: A; Day 19; Treatment: Tazemetostat with Fluconazole; Analyte: EPZ-6930 (ER-897387) | 2.02 (0.86)
  Part: A; Day 15; Treatment: Tazemetostat Alone; Analyte: EPZ006931 | 2.01 (0.89)
  Part: A; Day 19; Treatment: Tazemetostat with Fluconazole; Analyte: EPZ006931 | 2.47 (0.9)
  Part: A; Day 15; Treatment: Tazemetostat Alone; Analyte: EPZ034163 | 2.02 (1.26)
  Part: A; Day 19; Treatment: Tazemetostat with Fluconazole; Analyte: EPZ034163 | 2.02 (1.27)

15. Secondary Outcome: Part A: t1/2 of Tazemetostat Metabolites After Administration Alone and With Fluconazole
Time Frame: Days 15 and 19, 0 to 8 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: hours
Arm/Group | Part A
Number analyzed (Participants) | 14
hours
  Part: A; Day 15; Treatment: Tazemetostat Alone; Analyte: EPZ-6930 (ER-897387) | 2.89 (0.358)
  Part: A; Day 19; Treatment: Tazemetostat with Fluconazole; Analyte: EPZ-6930 (ER-897387) | 3.92 (0.621)
  Part: A; Day 15; Treatment: Tazemetostat Alone; Analyte: EPZ006931 | 3.24 (0.565)

16. Secondary Outcome: Part A: Exposure of Fluconazole After Administration of 400 mg Once Daily for 4 Days (AUC0-8)
Time Frame: Day 19, 0 to 8 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part A
Number analyzed (Participants) | 14
h*ng/mL | 170000 (48300)

17. Secondary Outcome: Part A: Cmax of Fluconazole After Administration of 400mg Once Daily for 4 Days
Time Frame: Day 19, 0 to 8 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A
Number analyzed (Participants) | 14
ng/mL | 25900 (6500)

18. Secondary Outcome: Part A: Tmax of Fluconazole After Administration of 400mg Once Daily for 4 Days
Time Frame: Day 19, 0 to 8 hours post-dose
Measure: Median (Standard Deviation); unit: hours
Arm/Group | Part A
Number analyzed (Participants) | 14
hours | 1.48 (1.95)

19. Secondary Outcome: The Antitumor Activity of Tazemetostat Will be Assessed in Patients With Diffuse Large B-cell Lymphoma (DLBCL), Marginal Zone Lymphoma (MZL), Follicular Lymphoma (FL) or Advanced Solid Tumors .
Description: Objective response rate (ORR: complete response [CR] or PR) and disease control rate (DCR: CR or PR, or stable disease lasting 24 weeks or longer from start of treatment with tazemetostat) using Lugano Classification for subjects with lymphoma, or Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 for subjects with solid tumors.
Time Frame: Within 28 days of Day 1, 8 weeks, 16 weeks, 24 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Lymphoma: Subjects with B-cell lymphomas
- Advanced Solid Tumors: Subjects with Advanced Solid Tumors
Arm/Group | Lymphoma | Advanced Solid Tumors
Number analyzed (Participants) | 13 | 16
Participants
  Complete response (CR) | 1 | 0
  Partial response (PR) | 1 | 2
  Stable disease (SD) | 0 | 9
  Progressive disease (PD) | 2 | 5
  Not evaluable, missing, or unknown | 9 | 3
  Objective Response Rate (ORR) | 2 | 2
  Disease control rate (DCR) at 24 weeks | 2 | 4
  Number of responders (achieving a CR or PR) | 2 | 2

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over a period of 2 years.
Arm/Group | Part A | Part B
All-Cause Mortality (participants affected / at risk) | 1/16 | 3/16
Serious Adverse Events (participants affected / at risk) | 4/16 | 6/16
Other Adverse Events (participants affected / at risk) | 12/16 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A (N=16) | Part B (N=16)
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A (N=16) | Part B (N=16)
Nausea (Gastrointestinal disorders) | 6 | 3
Diarrhoea (Gastrointestinal disorders) | 4 | 4
Vomiting (Gastrointestinal disorders) | 4 | 3
Flatulence (Gastrointestinal disorders) | 2 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 4
Eructation (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 6 | 8
Asthenia (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Face oedema (General disorders) | 0 | 1
Generalised oedema (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Dizziness (Nervous system disorders) | 3 | 0
Dysgeusia (Nervous system disorders) | 2 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Brain compression (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Fungal skin infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2
Viral rash (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Otitis media bacterial (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 0
Ocular discomfort (Eye disorders) | 1 | 0
Photophobia (Eye disorders) | 1 | 0
Macular oedema (Eye disorders) | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 0 | 2
Insomnia (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood calcium decreased (Investigations) | 0 | 1
Blood immunoglobulin G decreased (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 2
Testicular swelling (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Hot flush (Vascular disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT03028103/Prot_SAP_000.pdf